CLINICAL TRIAL: NCT04389515
Title: Evaluation of Pregnant Women Diagnosed With COVID-19 With "Post-operative Recovery Index" and "Prenatal Care Satisfaction and Patient Expectations Scale"
Brief Title: Postoperative Recovery Index, Patient Expectations and Satisfaction With Prenatal Care Instrument in Pregnant Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Aldikactioglu Talmac, MD, Specialist of Obstetrics and Gynecology, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: MTalmac3
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Prenatal Care; Postoperative Care
Keywords: COVID-19; Prenatal Care; Postoperative Care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to provide optimum care to postoperative patients diagnosed with COVID-19 (after cesarean) and to help them with recovery, to determine and assist the expectation and satisfaction of pregnant women with COVID-19 regarding prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with COVID-19

Exclusion Criteria:

* Patient giving Preterm Labor

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: As the patient group, two groups of 75 persons, each of whom are between the ages of 18-45 and who are diagnosed with COVID-19 in reproductive age and healthy pregnant women, will be selected. Patients diagnosed with COVID-19 giving birth with cesarean at term and patients who are followed up with COVID-19 diagnosis before the prenatal period will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-09-25 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pregnant women diagnosed with COVID-19 with "Post-operative Recovery Index" and "Prenatal Care Satisfaction and Patient Expectations Scale" | 3 Months
  The benefit we expect from the study is to be able to provide optimum care to postoperative patients (after cesarean) diagnosed with COVID-19 and to help them with recovery, to identify and assist the expectation and satisfaction of pregnant women with COVID-19 regarding prenatal care.

SECONDARY OUTCOMES:
Evaluation of pregnant women diagnosed with COVID-19 with "Post-operative Recovery Index" and "Prenatal Care Satisfaction and Patient Expectations Scale" | 3 Months
  To determine the differences between healthy pregnant women in the control group and pregnant women diagnosed with COVID-19 in the study group in terms of postoperative care and prenatal care expectations.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Halkali, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Omar MA, Schiffman RF, Bingham CR. Development and testing of the patient expectations and satisfaction with prenatal care instrument. Res Nurs Health. 2001 Jun;24(3):218-29. doi: 10.1002/nur.1024. PMID 11526620
- [Background] Cengiz H, Aygin D. Validity and reliability study of the Turkish version of the Postoperative Recovery Index of patients undergoing surgical intervention. Turk J Med Sci. 2019 Apr 18;49(2):566-573. doi: 10.3906/sag-1806-33. PMID 30893985